CLINICAL TRIAL: NCT05875883
Title: Anatomical Landmarks for Identifying the Phrenic Nerve With Ultrasound in Intensive Care Unit
Brief Title: Phrenic Identification in the ICU
Status: Active, not recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 23-083
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Ventilator Lung; Ventilator-Induced Lung Injury; Diaphragm Disease; Phrenic Nerve; Phrenic Nerve Stimulation; Neck Anatomy; Ultrasound
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Neck ultrasound — The investigators will scan patients' necks with an ultrasound and look for anatomical landmarks to identify the phrenic nerve

SUMMARY:
This will be a prospective observational study where the investigator will scan patients' necks with an ultrasound and look for anatomical landmarks that may help identify the phrenic nerve.

DETAILED DESCRIPTION:
Patients under protective mechanical ventilation, an intervention that saves lives, may need sedation and paralyzing agents. However, sedation and paralyzing agents are associated with multiple complications, including diaphragm dysfunction.

Several strategies have been proposed to reduce diaphram dysfunction. A novel approach is to stimulate the phrenic nerve, either transvenously or transcutaneously. Transvenous stimulation requires a catheter, which eventually is associated with increased risk of infection and thrombosis. In this scenario, transcutaneous phrenic nerve pacing is attractive but may be more susceptible to patients' anthropometric measures.

The correlation between patients' anthropometric measures and the location of the phrenic has been poorly studied.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Admitted to ICU

Exclusion Criteria

* Patients with a cervical spine collar
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2024-04-21 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the number of participants where the investigators will successfully identify the phrenic nerve using only ultrasound and anatomical landmarks | 25-30 minutes
To measure both phrenic nerves depth with an ultrasound in a heterogeneous population in the ICU | 25-30 minutes
To measure the distance, in milimeters, between each phrenic nerve and other homolateral cervical structures such as the carotid artery and the jugular vein | 25-30 minutes

SECONDARY OUTCOMES:
To describe potential clinical and anthropometric variables associated with phrenic nerve depth | 25-30 minutes
To assess how long it takes to find the phrenic nerve with ultrasound visualization. | 25-30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Reynolds SC, Meyyappan R, Thakkar V, Tran BD, Nolette MA, Sadarangani G, Sandoval RA, Bruulsema L, Hannigan B, Li JW, Rohrs E, Zurba J, Hoffer JA. Mitigation of Ventilator-induced Diaphragm Atrophy by Transvenous Phrenic Nerve Stimulation. Am J Respir Crit Care Med. 2017 Feb 1;195(3):339-348. doi: 10.1164/rccm.201502-0363OC. PMID 27500981
- [Background] Dres M, de Abreu MG, Merdji H, Muller-Redetzky H, Dellweg D, Randerath WJ, Mortaza S, Jung B, Bruells C, Moerer O, Scharffenberg M, Jaber S, Besset S, Bitter T, Geise A, Heine A, Malfertheiner MV, Kortgen A, Benzaquen J, Nelson T, Uhrig A, Moenig O, Meziani F, Demoule A, Similowski T; RESCUE-2 Study Group Investigators. Randomized Clinical Study of Temporary Transvenous Phrenic Nerve Stimulation in Difficult-to-Wean Patients. Am J Respir Crit Care Med. 2022 May 15;205(10):1169-1178. doi: 10.1164/rccm.202107-1709OC. PMID 35108175